CLINICAL TRIAL: NCT05667948
Title: Molecular Landscape Analysis and Treatment Options for Thymic Epithelial Tumors
Brief Title: Molecular Analysis and Treatment Options of Thymic Malignancies
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC002
Record Dates: First submitted 2022-11-30; First posted 2022-12-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Thymic Epithelial Tumor; Thymic Carcinoma; Thymic Cancer
Keywords: thymic malignancy; thymoma; chemotherapy; targeted therapy; immunotherapy; molecular landscape
MeSH Terms: conditions — Thymic epithelial tumor; Thymoma; Thymus Neoplasms | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimens are stored in the refrigerator at -20°C or -80°C as specified in the clinical trial protocol. Test specimens and backup specimens should be kept in separate refrigerators to prevent malfunction of one of the refrigerators. Centrifugation time, specimen collection and specimen storage time should be carried out in strict accordance with the requirements of the clinical trial protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chemotherapy — different treatments based on the molecular analysis
  Other Names: targeted therapy; immunotherapy

SUMMARY:
Thymic malignancies are the most common tumors of the anterior mediastinum, though surgery and radiation often effectively treat thymic carcinomas, a minority continue to progress and eventually lead to death. Therefore, there is an unmet need for more effective therapies for thymic malignancies. Considering the role of molecular alterations has yet to be defined in the treatment of thymoma and thymic malignancies, there is an urgent recognition that molecular alterations in the thymic malignancies are important to predict response and survival for novel targeted therapies.

In summary, identification of genetic alterations in thymic malignancies is increasingly essential to perform molecular diagnostics and individualized treatments. This project aims to create a registry of patients with thymic malignancies to further the characterization of molecular alterations and develop (novel) treatments based on the detection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of thymic malignancies
* 18 years of age or older
* Ability to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with thymic malignancies are with the standard treatment and/or are enrolled in the clinical trials.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 20 years
  Collect detailed clinical information on patients with thymic malignancies via the electronic medical records
Disease control rate (DCR) | 20 years
  Collect detailed clinical information on patients with thymic malignancies via the electronic medical records
Progression-free survival (PFS) | 20 years
  Collect detailed clinical information on patients with thymic malignancies via the electronic medical records

SECONDARY OUTCOMES:
Overall survival (OS) | 20 years
  Collect detailed clinical information on patients with thymic malignancies via the electronic medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaomin Niu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided